CLINICAL TRIAL: NCT01104272
Title: An Evaluation of the Treatment of Adipose Tissue Using a Focused Ultrasound Device in Subjects With Fitzpatrick IV-VI Skin Types
Brief Title: Subcutaneous Contouring Using High Intensity Focused Ultrasound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medicis Technologies Corporation (Industry)
Responsible Party: Patrick Martin, Executive Director, Clinical Affairs, Medicis Technologies Corporation
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: LP-1100-05
Record Dates: First submitted 2010-04-09; First posted 2010-04-15 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2011-01

CONDITIONS: Body Sculpting
Keywords: Ultrasound Treatment of Subcutaneous Adipose Tissue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Energy Level 1 (Experimental): Subcutaneous Adipose Tissue Treated With Energy Level 1.
  Interventions: Device: LipoSonix (Ultrasound treatment of Subcutaneous Adipose Tissue)

INTERVENTIONS:
Device: LipoSonix (Ultrasound treatment of Subcutaneous Adipose Tissue) — Study of Adipose Tissue Treatment Using Focused Ultrasound

SUMMARY:
The device delivers High Intensity Focused Ultrasound (HIFU) energy that can disrupt subcutaneous adipose tissue (SAT) to provide a non-invasive approach to body sculpting, such as a reduction in waist circumference.

ELIGIBILITY:
Inclusion Criteria:

All of the following inclusion criteria must be met at the time of screening before the subject is enrolled into the study:

1. Male or female subjects, 18 to 65 years of age
2. Body Mass Index ≤30
3. Thickness of subcutaneous adipose tissue in the anticipated treatment area of ≥ 2.5 cm
4. Subjects must agree to not alter their normal and regular diet or exercise routines during the course of the study.
5. Subjects must be of African descent AND have Fitzpatrick skin types IV, V, or VI.

Exclusion Criteria:

A subject is ineligible to participate in this study if they meet any of the following exclusion criteria at screening:

1. Female subject who is pregnant (i.e., has a positive urine pregnancy test), is suspected to be pregnant, or is lactating or becomes pregnant during the course of the study. (NOTE: Females of childbearing potential must have a negative urine pregnancy test prior to enrollment in the study.)
2. Subjects diagnosed with coagulation disorders or are receiving anticoagulant therapy or medications or dietary supplements which impede coagulation or platelet aggregation.
3. Subject has diabetes or cardiovascular disease.
4. Subject has had any aesthetic procedure to the region to be treated.
5. Subject has systemic skin disease or skin disease in the areas to be treated.
6. Subject has any abnormality of the skin or soft tissues of the abdominal wall in the areas to be treated.
7. Subject has had previous open or laparoscopic surgery in the anticipated treatment area.
8. Subjects is on prescription or over the counter weight reduction medication or programs, or had weight reduction procedures (e.g.: gastric bypass, Lap-Band, etc.)
9. Subject has skin or superficial tissue that does not lie flat on its own when the subject is in the supine position.
10. Subjects undergoing chronic steroid or immunosuppressive therapy.
11. Subjects who have cardiac pacemakers or any implantable electrical device, e.g. pacemaker, defibrillator, or neurostimulators.
12. Subjects who have metal implants of any type in the area to be treated.
13. History of cancer.
14. Subjects who have sensory loss or dysesthesia in the area to be treated.
15. Subject currently uses illicit drug(s) or abuses alcohol (defined as regular or daily consumption of more than 4 alcoholic drinks per day).
16. Subjects who cannot adhere to the study visit schedule (e.g., subjects not likely to stay in the study for a maximum of 27 weeks - screening through exit visit).
17. Subjects who are unable, or lack the capacity, to self consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in waist circumference | 12 weeks

SECONDARY OUTCOMES:
The change from Baseline in waist circumference measured after treatment, for the average of the two waist circumference measurements at the iliac crest as well as for each of the individual measurements. | 4 weeks
The change from Baseline in waist circumference measured after treatment, for the average of the two waist circumference measurements at the iliac crest as well as for each of the individual measurements. | 8 weeks
Patient satisfaction as recorded on the Subject Satisfaction Survey after treatment. | 1 week
Patient satisfaction as recorded on the Subject Satisfaction Survey after treatment. | 4 weeks
Patient satisfaction as recorded on the Subject Satisfaction Survey after treatment. | 8 weeks
Patient satisfaction as recorded on the Subject Satisfaction Survey after treatment. | 12 weeks
Visual Analog Scale (VAS) diary to record post treatment discomfort. | 1 week
Improvement as determined by a Global Aesthetic Improvement Scale (GAIS) score of 'improved' or 'much improved' at each post-baseline visit, as assessed by the Investigator. | 1 week
Improvement as determined by a Global Aesthetic Improvement Scale (GAIS) score of 'improved' or 'much improved' at each post-baseline visit, as assessed by the Investigator. | 4 weeks
Improvement as determined by a Global Aesthetic Improvement Scale (GAIS) score of 'improved' or 'much improved' at each post-baseline visit, as assessed by the Investigator. | 8 weeks
Improvement as determined by a Global Aesthetic Improvement Scale (GAIS) score of 'improved' or 'much improved' at each post-baseline visit, as assessed by the Investigator. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nowell Solish, MD, Principal Investigator — Dr. Nowell Solish Private Office; Sheetal Sapra, MD, Principal Investigator — Institute of Cosmetic and Laser Surgery
Locations (2):
- Canada (2):
  - Institute of Cosmetic and Laser Surgery, Oakville, Ontario
  - Dr. Nowell Solish Private Office, Toronto, Ontario